CLINICAL TRIAL: NCT04892030
Title: A Pilot Study of a Novel Ad Libitum Plant-Based Behavioral Weight Loss Treatment
Brief Title: Evaluating a Remotely Delivered Plant-Based Behavioral Weight Loss Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Evan Forman, Professor of Psychology, Drexel University, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EATVEG838
Record Dates: First submitted 2021-05-06; First posted 2021-05-19 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Overweight
Keywords: Weight loss; Behavioral weight loss; Overweight and obesity; Plant-based; Lifestyle modification
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will be prescribed a non-energy-restricted whole food plant-based diet and will learn behavioral weight loss strategies remotely, through an e-learning platform.
  Interventions: Behavioral: Whole Food Plant-Based Behavioral Weight Loss Treatment

INTERVENTIONS:
Behavioral: Whole Food Plant-Based Behavioral Weight Loss Treatment — Over the course of 12-weeks, participants will be prescribed a non-energy-restricted whole food plant-based diet and will learn behavioral weight loss strategies through an e-learning platform. Each week, participants will also complete a 15-minute coaching call to provide positive reinforcement and problem-solving support.

SUMMARY:
Many individuals do not achieve clinically significant weight loss following traditional lifestyle modification interventions, potentially because weight loss is dependent upon calorie tracking compliance (to achieve calorie prescriptions), which decreases over time for most. By contrast, non-energy-restricted whole food plant-based diets (WFPBD) have been demonstrated to promote clinically significant weight loss even without calorie prescriptions. The present pilot trial represents the first, to the knowledge of our study team, to empirically test a remotely delivered WFPBD behavioral weight loss intervention for adults with overweight or obesity. Over 12-weeks, participants (N = 21) will follow a non-energy-restricted WFPBD and received nutritional counseling and behavioral weight loss intervention. Participation will occur in two phases (Phase 1: n = 7; Phase 2: n = 14), between which iterative changes to the intervention will be made. Assessments will occur at baseline, mid-treatment, post-treatment, and 3-month follow-up. Data will be analyzed using an intent-to-treat approach. The primary aims of the study will be to assess retention feasibility and acceptability. The secondary aims will be to evaluate the preliminary effectiveness of the intervention on: (1) percent weight loss; (2) dietary intake (i.e., increased intake of low-fat plant-based whole foods and decreased in intake of processed foods and animal products); and (3) waist circumference. The exploratory aims will be to evaluate the preliminary effectiveness of the intervention on physical- and mental health-related quality of life, and to examine potential moderators of treatment success (plant-based diet history, internal disinhibition, social support vs. social sabotage, self-compassion, and psychological flexibility).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75
* Current BMI ≥ 25 kg/m2
* Reporting a desire to lose weight
* Have at-home internet access
* Proficiency in speaking, reading, and writing English
* Willing to consume a whole foods plant-based diet for the study duration

Exclusion Criteria:

* Use of medications for weight loss
* Recent weight loss (≥5% weight loss in prior 3-months)
* Current or planned pregnancy within the study period
* History of bariatric surgery
* Currently following a low-fat plant-based diet
* Diagnosis of a serious medical condition influencing weight, appetite, or eating behavior
* Diagnosis of a serious psychiatric condition that may influence weight, appetite, or eating behavior
* Current substance use disorder
* Participation in a concurrent weight loss program
* Planning on quitting smoking over the intervention period (if current smoker)
* Eating pathology (lifetime history of an eating disorder, ≥ 9 binge eating episodes in the past 3 months, or > 5 compensatory episodes in the past 3 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Retention feasibility as assessed by the number of participants successfully retained in the intervention | Week 12 (post-intervention)
  The number of participants who are retained in the study, as defined by completing the post-treatment assessment and at least 10 out of 12 of the weekly intervention modules. Successful retention will be defined as at least 80% of participants being retained in the study.
Acceptability as assessed by self-reported acceptability of the intervention | Week 12 (post-intervention)
  Acceptability will be assessed with three items, in which participants will report the degree to which they were satisfied with the intervention, found the intervention to be helpful, and the likelihood that they would recommend it to family/friends on a Likert scale ranging from 1 (Not at all) to 5 (Very much).

SECONDARY OUTCOMES:
Preliminary effectiveness of the intervention on weight loss, as assessed by self-reported weight from baseline to post-intervention | Measured once weekly from Week 0 (baseline) to Week 12 (post-intervention), and at 3-month follow-up
  Weight loss will be self-reported by participants weekly, and at baseline, mid-treatment, post-treatment, and 3-month follow-up. To evaluate the preliminary effectiveness of the intervention on weight loss, percent weight change from baseline to post-intervention will be evaluated. Preliminary weight loss effectiveness will be defined as at least 50% of participants losing at least 5% of their initial body weight by post-treatment.
Preliminary effectiveness of the intervention on dietary intake, as assessed by self-reported dietary intake from baseline to post-intervention | Week 0 (baseline), Week 6 (mid-treatment), Week 12 (post-intervention), and 3-month follow-up
  Dietary intake will be assessed using a food frequency questionnaire tailored to examine adherence to the prescribed intervention (whole food plant-based) diet. A dietary adherence index ranging from 0 (no adherence) to 100 (complete adherence) will be created, and preliminary dietary change effectiveness will be defined as at least 80% of participants improved their dietary adherence score by at least 20% by post-treatment.
Preliminary effectiveness of the intervention on waist circumference, as assessed by self-reported waist circumference from baseline to post-intervention | Week 0 (baseline), Week 6 (mid-treatment), Week 12 (post-intervention), and 3-month follow-up
  Waist circumference will be self-reported by participants weekly, and at baseline, mid-treatment, post-treatment, and 3-month follow-up. To evaluate the preliminary effectiveness of the intervention on waist circumference, waist circumference change from baseline to post-intervention will be examined. Preliminary weight loss effectiveness will be defined as at least 50% of participants losing at least 5% of their initial waist circumference by post-treatment.

OTHER OUTCOMES:
Preliminary effectiveness of the intervention on quality of life, as assessed by self-reported quality of life from baseline to post-intervention | Week 0 (baseline), Week 6 (mid-treatment), Week 12 (post-intervention), and 3-month follow-up
  Quality of life will be assessed using the 36-item Short-Form General Health Survey (SF-36). The SF-36 assesses eight domains: physical functioning, limits due to physical health, pain, general health, energy/fatigue, social functioning, emotional wellbeing, and mental health. Scores in each domain are converted to a scale from 0 to 100, with higher scores indicating better functioning in each domain. This scale produces both physical and mental health component summaries, both of which will be examined. A reliable change index at the .20 level will be calculated for both the physical- and mental- health-related component scores. If the product exceeds a z-score of 1.282 at post-treatment, reflecting 80% confidence, then results will be defined as suggestive of preliminary quality of life effectiveness.
Association between plant-based diet history at Week 0 (baseline) and percent weight loss at Week 12 (post-treatment) | Week 0 (baseline) and Week 12 (post-treatment)
  To assess plant-based diet history, a plant-based diet familiarity score will be computed from participants' self-reported familiarity with plant-based diets, reported on a scale ranging from 0 (Not at all familiar) to 4 (Very familiar), and from reports of whether they have eaten a plant-based diet in the past, for at least 3-months. Participants will be given 4 points if previously vegan, 3 if previously vegetarian, 2 if previously pescatarian or 1 if previously semi-vegetarian ("flexitarian"). These scores will be added to self-reported plant-based diet familiarity, resulting in a "plant-based diet familiarity" score that could range from 0 to 7. To evaluate the potential moderating effect of plant-based diet history on weight loss outcomes, the correlation between plant-based diet history and post-treatment percent weight loss will be examined.
Association between social support vs. social sabotage at Week 6 (mid-treatment) and percent weight loss at Week 12 (post-treatment) | Week 6 (mid-treatment) and Week 12 (post-treatment)
  To assess social support vs. social sabotage, participants will complete the Social Support and Sabotage Scale from Ball & Crawford (2006). On this measure, participants separately rate the degree to which friends and family act in ways that support or hinder their healthy eating efforts with a Likert scale ranging from 1 (Almost never) to 5 (Almost always). Scores will be averaged for each subscale to compute: 1) support for health behaviors from friends, 2) support for health behaviors from family, 3) sabotage for health behaviors from friends, and 4) sabotage for health behaviors from family. To evaluate the potential moderating effect of social support vs. social sabotage on weight loss outcomes, the correlations between social support vs. social sabotage for health behavior scores and post-treatment percent weight loss will be examined.
Association between internal disinhibition at Week 0 (baseline) and percent weight loss at Week 12 (post-treatment) | Week 0 (baseline) and Week 12 (post-treatment)
  To assess internal disinhibition, participants will complete the disinhibition subscale from the Mindful Eating Questionnaire (MEQ; Framson et al., 2009). Responses are on a Likert scale ranging from 1 (Never/Rarely) to 4 (Usually/Always). Scores for each item are averaged to compute an overall disinhibition score. To evaluate the potential moderating effect of internal disinhibition on weight loss outcomes, the correlation between internal disinhibition and post-treatment percent weight loss will be examined.
Association between self-compassion at Week 0 (baseline) and percent weight loss at Week 12 (post-treatment) | Week 0 (baseline) and Week 12 (post-treatment)
  To assess self-compassion, participants will complete the Self-Compassion Scale-Short Form, which assess how participants generally treat themselves during difficult times. Responses are on a Likert scale ranging from 1 (Almost never) to 5 (Almost always). Scores for each item are averaged to compute an overall self-compassion score. To evaluate the potential moderating effect of self-compassion on weight loss outcomes, the correlation between self-compassion and post-treatment percent weight loss will be examined.
Association between psychological flexibility at Week 6 (mid-treatment) and percent weight loss at Week 12 (post-treatment) | Week 6 (mid-treatment) and Week 12 (post-treatment)
  To assess psychological flexibility, participants will complete the personalized psychological flexibility index, which assesses the ability to pursue valued life aims despite the presence of distress. Responses are on a Likert scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree). Scores for each item are averaged to compute an overall psychological flexibility score. To evaluate the potential moderating effect of psychological flexibility on weight loss outcomes, the correlation between psychological flexibility and post-treatment percent weight loss will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Forman, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Weight Eating and Lifestyle Science Center, Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in a public repository stripped of any identifying participant information.
Supporting Information: SAP, Analytic Code
Time Frame: Immediately following manuscript publication, the study data study and statistical code used for analyses will be shared.
URL: https://osf.io/mtp73/?view_only=0a0c51abcd7c45b0a6283d9c1d0fc50d

REFERENCES:
- [Derived] Chwyl C, Wright N, M Turner-McGrievy G, L Butryn M, M Forman E. Remotely Delivered Behavioral Weight Loss Intervention Using an Ad Libitum Plant-Based Diet: Pilot Acceptability, Feasibility, and Preliminary Results. JMIR Form Res. 2022 Jun 23;6(6):e37414. doi: 10.2196/37414. PMID 35737443